CLINICAL TRIAL: NCT05686200
Title: The Effect of Intelligent Forearm Isometric Exercise on Vascular Function, Hand Grip Strength and Adherence in Patients With First Autologous Arteriovenous Fistula After Surgery
Brief Title: The Effect of Intelligent Exercise on Vascular Function, Grip Strength and Adherence in Patients With AVF After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Taiwan Nurses Association (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, Ph.D., RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: NTUNHS-012
Record Dates: First submitted 2022-11-24; First posted 2023-01-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Arteriovenous Fistula; Isometric Exercise
Keywords: vascular function; muscle strength; adherence
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: Two-group Parallel Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants performed wrist-forearm exercise training within 2 weeks after the operation, that is, from 24 hours to 2 weeks after the operation, twice a day in the morning and evening, 3 groups each time, and each single item was repeated 5 times in each group (maintain for 5 seconds). Exercise for 40 minutes a day, use the mobile phone to install the forearm isometric exercise software program within the 3rd to 8th week, use the Bluetooth device to connect the hand-held gripper to perform the forearm isometric exercise, 2 times a day, morning and evening, and train 3 groups each time, 20 times each time , hand grip strength for 3 seconds each time, increase by 1 second per week, and rest for 90 seconds between groups.
  Interventions: Behavioral: Forearm isometric exercise intervention program
- Control group (Other): The control group began to use soft rubber balls for isometric contraction exercise from the 2nd day to the 8th week after operation. 2 times a day in the morning and evening, 3 groups of training each time, each group holds the ball for 5 minutes, and rests for 90 seconds between groups. Each grip training must be completed 20 times within 1 minute (keep 3 seconds each time in the first week) , increase by 2 seconds every week, and keep each grasping time for 10 seconds from the 5th to the 8th week.
  Interventions: Behavioral: Forearm isometric exercise intervention program

INTERVENTIONS:
Behavioral: Forearm isometric exercise intervention program — Experimental group using the intelligent gripper for forearm isometric exercise in the 3rd to 8th participants after operation, and using the smart mobile phone to install the forearm isometric exercise training game program software to provides an interactive and real- time exercise grip strength feedback mechanism, which are uses the interest of the participant to complete the forearm isometric exercise every day, and can implement the isometric exercise training for fistulization. Study nurses will track exercise adherence with telephone interviews 2, 4 and 8 participants after participant exercise intervention.

SUMMARY:
Isometric exercise can effectively promote the vascular function of arteriovenous fistula and increase hand grip strength, but patients needs to perform isometric exercises patiently. The purpose of this study want investigate the effect of using individual intelligent devices for forearm isometric exercise training on the increase of arteriovenous fistula vascular function and hand grip strength, and the improvement of patients' adherence with forearm isometric exercise.

DETAILED DESCRIPTION:
An arteriovenous fistula(AVF) is the most preferred and safe vascular access for long-term hemodialysis patients. Isometric exercise can effectively promote the vascular function of AVF and increase hand grip strength, but patients needs to perform isometric exercises patiently. However, the patient's disease factors, muscle soreness caused by the exercise process, etc., may easily prevent the patient from effectively performing isometric exercise every day.This study will be the first isometric exercise training intervention program for eight weeks after AVF surgery with an intelligent device in Taiwan. Investigators expect to promote the vascular function of AVF and increase hand grip strength, as well as improve participant' adherence performance after the re-intervention protocol. To construct an intelligent forearm isometric exercise, as a reference for clinical care guidance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* Regular follow-up in the nephrology clinic
* Diagnosed with chronic kidney disease at stage 5 (or 5D)
* Expect to do the first autologous arteriovenous fistula surgery

Exclusion Criteria:

* Not the first autologous arteriovenous fistula surgery
* Have undergone percutaneous transluminal angioplasty in the arm receiving autologous arteriovenous fistula
* Have undergone orthopedic disease-related surgery in the arm receiving autologous arteriovenous fistula
* Have been cardiovascular events within the past 3 months
* Have been heart function Left ventricular ejection fraction within the past 3 months <30%.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Vascular function in postoperative arteriovenous fistula | Baseline, pre-intervention (T0)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, professional radiology technicians used ultrasonic instruments to check and record the inner diameter of the blood vessel and the peak blood flow velocity of the drainage vein of the participant's arteriovenous fistula
Change from Baseline Vascular function in postoperative arteriovenous fistula at two weeks | Baseline and Weeks 2 (T1)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, professional radiology technicians used ultrasonic instruments to check and record the inner diameter of the blood vessel and the peak blood flow velocity of the drainage vein of the participant's arteriovenous fistula
Change from Baseline Vascular function in postoperative arteriovenous fistula at four weeks | Baseline and Weeks 4 (T2)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, professional radiology technicians used ultrasonic instruments to check and record the inner diameter of the blood vessel and the peak blood flow velocity of the drainage vein of the participant's arteriovenous fistula
Change from Baseline Vascular function in postoperative arteriovenous fistula at eight weeks | Baseline and Weeks 8 (T3)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, professional radiology technicians used ultrasonic instruments to check and record the inner diameter of the blood vessel and the peak blood flow velocity of the drainage vein of the participant's arteriovenous fistula
Clinical assessment of arteriovenous fistula maturity | Baseline, post-intervention(T1)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, senior hemodialysis nurses assessed whether there were palpable tremors in the blood vessels of the arteriovenous fistula, and whether there were obvious visible veins and arteriovenous in the arteriovenous fistula. Fistula with or without visible vessels >10 cm line.
Change from Baseline Clinical assessment of arteriovenous fistula maturity at four weeks | Baseline and Weeks 4(T2)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, senior hemodialysis nurses assessed whether there were palpable tremors in the blood vessels of the arteriovenous fistula, and whether there were obvious visible veins and arteriovenous in the arteriovenous fistula. Fistula with or without visible vessels >10 cm line.
Change from Baseline Clinical assessment of arteriovenous fistula maturity at eight weeks | Baseline and Weeks 8(T3)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, senior hemodialysis nurses assessed whether there were palpable tremors in the blood vessels of the arteriovenous fistula, and whether there were obvious visible veins and arteriovenous in the arteriovenous fistula. Fistula with or without visible vessels >10 cm line.
Ultrasonic evaluation of arteriovenous fistula maturity | Baseline, two weeks after intervention(T1)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, the vascular radiologist used the ultrasound equipment of the Philips ClearVue 550 ultrasound system (ClearVue 550, USA) to assess whether the participant's arteriovenous fistula was far from the skin. <6mm, whether the inner diameter of the outflow brachiocephalic vein is >6mm, whether the brachial artery flow rate is >600 mL/min, and record the measured values.
Change from Baseline Ultrasonic evaluation of arteriovenous fistula maturity at four weeks | Baseline and Weeks 4(T2)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, the vascular radiologist used the ultrasound equipment of the Philips ClearVue 550 ultrasound system (ClearVue 550, USA) to assess whether the participant's arteriovenous fistula was far from the skin. <6mm, whether the inner diameter of the outflow brachiocephalic vein is >6mm, whether the brachial artery flow rate is >600 mL/min, and record the measured values.
Change from Baseline Ultrasonic evaluation of arteriovenous fistula maturity at eight weeks | Baseline and Weeks 8(T3)
  After the participants rested for 5 minutes at the temperature of the ultrasound room set at 25°C, the vascular radiologist used the ultrasound equipment of the Philips ClearVue 550 ultrasound system (ClearVue 550, USA) to assess whether the participant's arteriovenous fistula was far from the skin. <6mm, whether the inner diameter of the outflow brachiocephalic vein is >6mm, whether the brachial artery flow rate is >600 mL/min, and record the measured values.
Hand Grip Strength | Baseline, before exercise intervention(T0)
  Grip Strength Assessment using a hydraulic hand-held dynamometer (Takei Hand Grip Dynamometer, Japan), the arm muscle strength of the participants in the non-dominant hand was assessed. The participants sits on a chair with a backrest, with the hips bent 90 degrees, feet flat on the ground, shoulders adducted, elbows bent 90 degrees, the non-dominant arm is in a neutral position, the wrist is maintained at an extension angle of 0-30 degrees, and the ulnar side is biased. Move 0~15 degrees. A total of three measurements will be taken with a one-minute rest in between, and measurements were made in kilograms (Kg). In addition, on the 15th day after the operation, the experimental group started to use the smart grip device for forearm isometric exercise and recorded the data after grip strength training.
Change from Baseline Hand Grip Strength at two weeks | Baseline and Weeks 2 (T1)
  Grip Strength Assessment using a hydraulic hand-held dynamometer (Takei Hand Grip Dynamometer, Japan), the arm muscle strength of the participants in the non-dominant hand was assessed. The participants sits on a chair with a backrest, with the hips bent 90 degrees, feet flat on the ground, shoulders adducted, elbows bent 90 degrees, the non-dominant arm is in a neutral position, the wrist is maintained at an extension angle of 0-30 degrees, and the ulnar side is biased. Move 0~15 degrees. A total of three measurements will be taken with a one-minute rest in between, and measurements were made in kilograms (Kg). In addition, on the 15th day after the operation, the experimental group started to use the smart grip device for forearm isometric exercise and recorded the data after grip strength training.
Change from Baseline Hand Grip Strength at four weeks | Baseline and Weeks 4(T2)
  Grip Strength Assessment using a hydraulic hand-held dynamometer (Takei Hand Grip Dynamometer, Japan), the arm muscle strength of the participants in the non-dominant hand was assessed. The participants sits on a chair with a backrest, with the hips bent 90 degrees, feet flat on the ground, shoulders adducted, elbows bent 90 degrees, the non-dominant arm is in a neutral position, the wrist is maintained at an extension angle of 0-30 degrees, and the ulnar side is biased. Move 0~15 degrees. A total of three measurements will be taken with a one-minute rest in between, and measurements were made in kilograms (Kg). In addition, on the 15th day after the operation, the experimental group started to use the smart grip device for forearm isometric exercise and recorded the data after grip strength training.
Change from Baseline Hand Grip Strength at eight weeks | Baseline and Weeks 8 (T3)
  Grip Strength Assessment using a hydraulic hand-held dynamometer (Takei Hand Grip Dynamometer, Japan), the arm muscle strength of the participants in the non-dominant hand was assessed. The participants sits on a chair with a backrest, with the hips bent 90 degrees, feet flat on the ground, shoulders adducted, elbows bent 90 degrees, the non-dominant arm is in a neutral position, the wrist is maintained at an extension angle of 0-30 degrees, and the ulnar side is biased. Move 0~15 degrees. A total of three measurements will be taken with a one-minute rest in between, and measurements were made in kilograms (Kg). In addition, on the 15th day after the operation, the experimental group started to use the smart grip device for forearm isometric exercise and recorded the data after grip strength training.

SECONDARY OUTCOMES:
Rate of participants' exercise adherence | Baseline, two weeks after intervention(T1)
  Participants began to self-register daily exercise times, each exercise group, each exercise frequency, and self-assessed daily exercise effort scores in the exercise log on the second day after the operation, and the end of the 8th week of exercise post-compute rate of adherence.
Change from Baseline Rate of Adherence at four weeks | Baseline and Weeks 4(T2)
  Participants began to self-register daily exercise times, each exercise group, each exercise frequency, and self-assessed daily exercise effort scores in the exercise log on the second day after the operation, and the end of the 8th week of exercise post-compute rate of adherence.
Change from Baseline Rate of Adherence at eight weeks | Baseline and Weeks 8(T3)
  Participants began to self-register daily exercise times, each exercise group, each exercise frequency, and self-assessed daily exercise effort scores in the exercise log on the second day after the operation, and the end of the 8th week of exercise post-compute rate of adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alikari V, Tsironi M, Matziou V, Tzavella F, Stathoulis J, Babatsikou F, Fradelos E, Zyga S. The impact of education on knowledge, adherence and quality of life among patients on haemodialysis. Qual Life Res. 2019 Jan;28(1):73-83. doi: 10.1007/s11136-018-1989-y. Epub 2018 Sep 3. PMID 30178430
- [Background] Andrade FP, Benvenutti H, da Silva KC, Rovedder PME. Effects of upper limb exercise programs on the arteriovenous fistula in patients on hemodialysis: A systematic review and meta-analysis. J Vasc Access. 2022 Sep;23(5):770-777. doi: 10.1177/11297298211001166. Epub 2021 Apr 27. PMID 33904355
- [Background] Bohannon RW. Muscle strength: clinical and prognostic value of hand-grip dynamometry. Curr Opin Clin Nutr Metab Care. 2015 Sep;18(5):465-70. doi: 10.1097/MCO.0000000000000202. PMID 26147527
- [Background] Collado-Mateo D, Lavin-Perez AM, Penacoba C, Del Coso J, Leyton-Roman M, Luque-Casado A, Gasque P, Fernandez-Del-Olmo MA, Amado-Alonso D. Key Factors Associated with Adherence to Physical Exercise in Patients with Chronic Diseases and Older Adults: An Umbrella Review. Int J Environ Res Public Health. 2021 Feb 19;18(4):2023. doi: 10.3390/ijerph18042023. PMID 33669679
- [Background] Cronin J, Lawton T, Harris N, Kilding A, McMaster DT. A Brief Review of Handgrip Strength and Sport Performance. J Strength Cond Res. 2017 Nov;31(11):3187-3217. doi: 10.1519/JSC.0000000000002149. PMID 28820854
- [Background] Fontsere N, Mestres G, Yugueros X, Lopez T, Yuguero A, Bermudez P, Gomez F, Riambau V, Maduell F, Campistol JM. Effect of a postoperative exercise program on arteriovenous fistula maturation: A randomized controlled trial. Hemodial Int. 2016 Apr;20(2):306-14. doi: 10.1111/hdi.12376. Epub 2015 Oct 20. PMID 26486682
- [Background] Hawley-Hague H, Horne M, Skelton DA, Todd C. Review of how we should define (and measure) adherence in studies examining older adults' participation in exercise classes. BMJ Open. 2016 Jun 23;6(6):e011560. doi: 10.1136/bmjopen-2016-011560. PMID 27338884
- [Background] Ibeas J, Roca-Tey R, Vallespin J, Moreno T, Monux G, Marti-Monros A, Del Pozo JL, Gruss E, Ramirez de Arellano M, Fontsere N, Arenas MD, Merino JL, Garcia-Revillo J, Caro P, Lopez-Espada C, Gimenez-Gaibar A, Fernandez-Lucas M, Valdes P, Fernandez-Quesada F, de la Fuente N, Hernan D, Arribas P, Sanchez de la Nieta MD, Martinez MT, Barba A; por el Grupo Espanol Multidisciplinar del Acceso Vascular (GEMAV). Spanish Clinical Guidelines on Vascular Access for Haemodialysis. Nefrologia. 2017 Nov;37 Suppl 1:1-191. doi: 10.1016/j.nefro.2017.11.004. English, Spanish. PMID 29248052
- [Background] Kumar A/L S Katheraveloo K, Suryani Safri L, Guo Hou L, Hafiz Maliki A, Md Idris MA, Harunarashid H. Effect of isometric handgrip exercise on the size of cephalic veins in patients with stage 3 and 4 chronic kidney disease: A randomized controlled trial. J Vasc Access. 2020 May;21(3):372-378. doi: 10.1177/1129729819879314. Epub 2019 Oct 4. PMID 31581898
- [Background] Kong S, Lee KS, Kim J, Jang SH. The effect of two different hand exercises on grip strength, forearm circumference, and vascular maturation in patients who underwent arteriovenous fistula surgery. Ann Rehabil Med. 2014 Oct;38(5):648-57. doi: 10.5535/arm.2014.38.5.648. Epub 2014 Oct 30. PMID 25379494
- [Background] Lok CE, Huber TS, Lee T, Shenoy S, Yevzlin AS, Abreo K, Allon M, Asif A, Astor BC, Glickman MH, Graham J, Moist LM, Rajan DK, Roberts C, Vachharajani TJ, Valentini RP; National Kidney Foundation. KDOQI Clinical Practice Guideline for Vascular Access: 2019 Update. Am J Kidney Dis. 2020 Apr;75(4 Suppl 2):S1-S164. doi: 10.1053/j.ajkd.2019.12.001. Epub 2020 Mar 12. PMID 32778223
- [Background] Nantakool S, Srisuwan T, Reanpang T, Rerkasem K, Prasannarong M. A randomized controlled trial of the effect of postoperative hand exercise training on arteriovenous fistula maturation in patients with chronic kidney disease. J Vasc Surg. 2022 Jan;75(1):230-237. doi: 10.1016/j.jvs.2021.07.124. Epub 2021 Jul 24. PMID 34314831
- [Background] Oprea A, Molnar A, Vladutiu D, Scridon T, Trifan C, Sacui D, Sasarman V, Mircea PA. Correlation between preoperative vein and artery diameters and arteriovenous fistula outcome in patients with end-stage renal disease. Clujul Med. 2018 Oct;91(4):399-407. doi: 10.15386/cjmed-1080. Epub 2018 Oct 30. PMID 30564015
- [Background] Rothuizen TC, Wong C, Quax PH, van Zonneveld AJ, Rabelink TJ, Rotmans JI. Arteriovenous access failure: more than just intimal hyperplasia? Nephrol Dial Transplant. 2013 May;28(5):1085-92. doi: 10.1093/ndt/gft068. Epub 2013 Mar 29. PMID 23543595
- [Background] Salimi F, Majd Nassiri G, Moradi M, Keshavarzian A, Farajzadegan Z, Saleki M, Nikpoor A, Ghane M. Assessment of effects of upper extremity exercise with arm tourniquet on maturity of arteriovenous fistula in hemodialysis patients. J Vasc Access. 2013 Jul-Sep;14(3):239-44. doi: 10.5301/jva.5000123. Epub 2013 Jan 3. PMID 23283645
- [Background] Schmidli J, Widmer MK, Basile C, de Donato G, Gallieni M, Gibbons CP, Haage P, Hamilton G, Hedin U, Kamper L, Lazarides MK, Lindsey B, Mestres G, Pegoraro M, Roy J, Setacci C, Shemesh D, Tordoir JHM, van Loon M, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Lindholt J, Naylor R, Vega de Ceniga M, Vermassen F, Verzini F, Esvs Guidelines Reviewers, Mohaupt M, Ricco JB, Roca-Tey R. Editor's Choice - Vascular Access: 2018 Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Jun;55(6):757-818. doi: 10.1016/j.ejvs.2018.02.001. Epub 2018 May 2. No abstract available. PMID 29730128
- [Background] Silva IB, Barbosa JBN, Araujo AXP, Marinho PEM. Effect of an exercise program with blood flow restriction on the muscular strength of patients with chronic kidney disease: A randomized clinical trial. J Bodyw Mov Ther. 2021 Oct;28:187-192. doi: 10.1016/j.jbmt.2021.06.022. Epub 2021 Jun 23. PMID 34776140
- [Background] Sidawy AN, Gray R, Besarab A, Henry M, Ascher E, Silva M Jr, Miller A, Scher L, Trerotola S, Gregory RT, Rutherford RB, Kent KC. Recommended standards for reports dealing with arteriovenous hemodialysis accesses. J Vasc Surg. 2002 Mar;35(3):603-10. doi: 10.1067/mva.2002.122025. PMID 11877717
- [Background] Smith GE, Gohil R, Chetter IC. Factors affecting the patency of arteriovenous fistulas for dialysis access. J Vasc Surg. 2012 Mar;55(3):849-55. doi: 10.1016/j.jvs.2011.07.095. Epub 2011 Nov 8. PMID 22070937
- [Background] Tapia Gonzalez I, Esteve Simo V, Ibanez S, Moreno Guzman F, Fulquet Nicolas M, Duarte Gallego V, Saurina Sole A, Pou Potau M, Yeste Campos M, de Arellano Serna MR. Elderly patients, isometric exercise, and native vascular access maturation: An unsolved question? Hemodial Int. 2021 Apr;25(2):154-163. doi: 10.1111/hdi.12900. Epub 2020 Nov 5. PMID 33155357
- [Background] Hart A, Lentine KL, Smith JM, Miller JM, Skeans MA, Prentice M, Robinson A, Foutz J, Booker SE, Israni AK, Hirose R, Snyder JJ. OPTN/SRTR 2019 Annual Data Report: Kidney. Am J Transplant. 2021 Feb;21 Suppl 2:21-137. doi: 10.1111/ajt.16502. PMID 33595191
- [Background] Wilschut ED, Rotmans JI, Bos EJ, van Zoest D, Eefting D, Hamming JF, van der Bogt KEA. Supervised preoperative forearm exercise to increase blood vessel diameter in patients requiring an arteriovenous access for hemodialysis: rationale and design of the PINCH trial. J Vasc Access. 2018 Jan;19(1):84-88. doi: 10.5301/jva.5000826. PMID 29148008
- [Background] Hsiao YH, Shin ML, Huang CP, Chen SJ, Huang TY. [Using Interdisciplinary Cooperation to Improve the Rate of Proper Performance of a Hand Exercise Among Hemodialysis Patients With Arteriovenous Fistula Construction]. Hu Li Za Zhi. 2017 Jun;64(3):74-81. doi: 10.6224/JN.000042. Chinese. PMID 28580561
- [Background] Chen YC, Chang P. [Using eHealth in the Continuity Care of Chronic Kidney Disease: Opportunities and Considerations]. Hu Li Za Zhi. 2016 Apr;63(2):12-8. doi: 10.6224/JN.63.2.12. Chinese. PMID 27026552